CLINICAL TRIAL: NCT02189252
Title: A Randomized, Open-Label Crossover Study to Compare the Relative Bioavailability, Efficacy, and Safety of Epanova® and Lovaza® in Men and Women With a History of Pancreatitis
Brief Title: An Open-Label Crossover Study to Compare the Relative Bioavailability, Efficacy and Safety of Epanova® and Lovaza® in Men and Women With a History of Pancreatitis
Acronym: ECLIPSEIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D5880C00003; OM-EPA-013 (Other: Omthera)
Record Dates: First submitted 2014-06-23; First posted 2014-07-14 (Estimated); Results first posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-05

CONDITIONS: Severe Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- E4:L4 (Active Comparator): Crossover Sequence
  Interventions: Drug: Epanova; Drug: Lovaza
- L4:E4 (Active Comparator): Crossover Sequence
  Interventions: Drug: Epanova; Drug: Lovaza
- E2:L4 (Active Comparator): Crossover Sequence
  Interventions: Drug: Epanova; Drug: Lovaza
- L4:E2 (Active Comparator): Crossover Sequence
  Interventions: Drug: Epanova; Drug: Lovaza

INTERVENTIONS:
Drug: Epanova
Drug: Lovaza

SUMMARY:
This is a randomized, open-label crossover study. The primary objective of this study is to compare the relative bioavailability of eicosapentaenoic acid (EPA), docosahexaenoic acid (DHA), docosapentaenoic acid (DPA), and the ethyl esters of EPA and DHA in plasma from a single 2 g or 4 g dose of Epanova® or 4 g Lovaza®.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥18 years of age;
2. History of serum TG concentration ≥500 mg/dL within the past 5 years;
3. Have at least one episode of documented hospitalization for pancreatitis due to hypertriglyceridemia in his/her lifetime;
4. Have no health conditions that would prevent him/her from fulfilling the study requirements as judged by the Investigator on the basis of physical examination, ECG, medical history, and routine laboratory test results;
5. Willing to maintain his/her current activity level and to follow either the NCEP TLC diet with a caloric target for weight maintenance or a prescribed low-fat diet during the screening, treatment, and washout periods (Visits 1 through 6b; Weeks -4 through 12);
6. Willing to eat the standardized breakfast, lunch, and dinner meals and snacks before and during Visits 4b and 6b (Weeks 4 and 12);
7. Willing to abstain from alcohol consumption and avoid vigorous physical activity for 48 hours prior to Visits 3 through 6b (Weeks 0 through 12); and
8. Subject understands the study procedures and is willing and able to sign the informed consent form to participate in the study and the Health Insurance Portability and Accountability Act authorization for release of relevant protected health information to the Investigators and study personnel.

Exclusion Criteria:

1. An allergy or intolerance to omega-3 fatty acids, omega-3-acid ethyl esters, fish, or any of the components of the standardized breakfast, lunch, or dinner meals or snacks (as described to them by study staff)
2. Poorly controlled hypertension (resting blood pressure ≥160 mmHg systolic and/or ≥100 mmHg diastolic) prior to randomization (Visit 3 [Week 0])
3. A history of cancer (other than basal cell carcinoma) in the last 2 years
4. A recent cardiovascular event (i.e., myocardial infarction, acute coronary syndrome, new onset angina, stroke, transient ischemic attack, unstable congestive heart failure requiring a change in treatment), aortic aneurysm or resection, carotid endarterectomy, or revascularization procedure within the 6 months prior to Visit 1

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Lawless, MD, Principal Investigator — Biofortis, Inc Addison IL 60101
Locations (4):
- United States (3):
  - Research Site, Kansas City, Kansas
  - Research Site, Cincinnati, Ohio
  - Research Site, Philadelphia, Pennsylvania
- Research Site, Chocoutimi, Quebec, Canada

REFERENCES:
- [Derived] Dunbar RL, Gaudet D, Davidson M, Rensfeldt M, Yang H, Nilsson C, Kvarnstrom M, Oscarsson J. Omega-3 fatty acid exposure with a low-fat diet in patients with past hypertriglyceridemia-induced acute pancreatitis; an exploratory, randomized, open-label crossover study. Lipids Health Dis. 2020 May 30;19(1):117. doi: 10.1186/s12944-020-01295-7. PMID 32473640

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study subjects were recruited at 6 sites. In total, 30 subjects were screened, of which 15 were randomized to 1 of 4 treatment sequences.
Pre-assignment Details: No applicable
Groups:
- Treatment Sequence 1: Epanova 4g per day: Lovaza 4g per day
- Treatment Sequence 2: Lovaza 4 g per day:Epanova 4 g per day : 4 subjects
- Treatment Sequence 3: Epanova 2g per day:Lovaza 4g per day:
- Treatment Sequence 4: Lovaza 4g per day:Epanova 2g per day:
Period: Period 1 (Visit 4b, Week 4)
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4
Started | 4 | 4 | 3 | 4
Completed | 4 | 2 | 3 | 4
Not Completed | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Period 2 (Visit6b, Week 12)
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4
Started | 4 | 2 | 3 | 4
Completed | 4 | 2 | 3 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Sequence 1: Epanova 4 g per day:Lovaza 4 g per day
- Treatment Sequence 3: Epanova 2 g per day:Lovaza 4 g per day
- Treatment Sequence 4: Lovaza 4 g per day:Epanova 2 g per day: 4 subjects
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Total
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (6.86) | 46.0 (13.09) | 53.0 (16.46) | 53.5 (11.27) | 49.8 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 0 | 5
  Male | 3 | 1 | 2 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Baseline-adjusted AUC0-24 for Plasma Total EPA + Total DHA
Description: AUC0-24: Area under the plasma concentration versus time curve, from time 0 to 24 hours after start of the meal
Time Frame: participants were followed for the duration of study, up to 12 weeks, each treatment having a 4-week duration and a 4-week wash off period in between.
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nmol/mL
Groups:
- Epanova 2 g; Epanova 4 g; Lovaza 4 g: Once daily (QD)
Arm/Group | Epanova 2 g | Epanova 4 g | Lovaza 4 g
Number analyzed (Participants) | 6 | 6 | 12
hr*nmol/mL | 17000 (121.7) | 18000 (104.6) | 12500 (80.0)
Statistical Analysis 1: Comparison: Epanova 4 g vs Lovaza 4 g; In order to address the issue of multiple testing while maintaining overall type I error, a closed testing sequence was used involving 4 analyses stated in the primary objective of this study. In total, 4 statistical tests, each at a significance level of 5%, were carried along the fixed sequence until the first statistically non-significant treatment difference was observed (i.e. p-value>0.05). This is the first test in the fixed testing sequence; Test type: Superiority or Other; p = 0.2702, Mixed Models Analysis — The closed sequential testing procedure stopped at this step as the P Value is greater than 0.05; Geometric mean ratio in % = 160.05, 95% CI 2-sided [64.71 to 395.82]
Statistical Analysis 2: Comparison: Epanova 2 g vs Lovaza 4 g; In order to address the issue of multiple testing while maintaining overall type I error, a closed testing sequence was used involving 4 analyses stated in the primary objective of this study. In total, 4 statistical tests, each at a significance level of 5%, were carried along the fixed sequence until the first statistically non-significant treatment difference was observed (i.e. p-value>0.05). This is the second test in the fixed testing sequence; Test type: Superiority or Other; p = 0.6367, Mixed Models Analysis — The p-value was only interpreted descriptively; Geometric mean ratio in % = 121.61, 95% CI 2-sided [49.17 to 300.76]

2. Primary Outcome: Baseline-adjusted Cmax for Plasma Total EPA + Total DHA
Description: Cmax: Maximum measured plasma concentration over the time span specified
Time Frame: as for outcome 1
Population: PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/mL
Arm/Group | Epanova 2 g | Epanova 4 g | Lovaza 4 g
Number analyzed (Participants) | 6 | 6 | 12
nmol/mL | 1090 (78.6) | 1200 (70.2) | 712 (76.7)
Statistical Analysis 1: Comparison: Epanova 4 g vs Lovaza 4 g; In order to address the issue of multiple testing while maintaining overall type I error, a closed testing sequence was used involving 4 analyses stated in the primary objective of this study. In total, 4 statistical tests, each at a significance level of 5%, were carried along the fixed sequence until the first statistically non-significant treatment difference was observed (i.e. p-value>0.05). This is the third test in the fixed testing sequence; Test type: Superiority or Other; p = 0.0511, Mixed Models Analysis — The p-value was only interpreted descriptively; Geometric mean ratio in % = 193.91, 95% CI 2-sided [99.61 to 377.47]
Statistical Analysis 2: Comparison: Epanova 2 g vs Lovaza 4 g; In order to address the issue of multiple testing while maintaining overall type I error, a closed testing sequence was used involving 4 analyses stated in the primary objective of this study. In total, 4 statistical tests, each at a significance level of 5%, were carried along the fixed sequence until the first statistically non-significant treatment difference was observed (i.e. p-value>0.05). This is the fourth test in the fixed testing sequence; Test type: Superiority or Other; p = 0.3543, Mixed Models Analysis — The p-value was only interpreted descriptively; Geometric mean ratio in % = 133.32, 95% CI 2-sided [68.49 to 259.52]

3. Secondary Outcome: Baseline-adjusted AUC0-24 for Plasma Total EPA
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ug/mL
Arm/Group | Epanova 2 g | Epanova 4 g | Lovaza 4 g
Number analyzed (Participants) | 6 | 6 | 12
hr*ug/mL | 3510 (117.8) | 3930 (83.0) | 1730 (78.4)
Statistical Analysis 1: Comparison: Epanova 4 g vs Lovaza 4 g; Test type: Superiority or Other; p = 0.0210, Mixed Models Analysis; Geometric mean ratio in % = 259.19, 95% CI 2-sided [119.75 to 560.99]
Statistical Analysis 2: Comparison: Epanova 2 g vs Lovaza 4 g; Test type: Superiority or Other; p = 0.1256, Mixed Models Analysis; Geometric mean ratio in % = 177.95, 95% CI 2-sided [82.22 to 385.16]

4. Secondary Outcome: Baseline-adjusted Cmax for Plasma Total EPA
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Epanova 2 g | Epanova 4 g | Lovaza 4 g
Number analyzed (Participants) | 6 | 6 | 12
ug/mL | 221 (83.0) | 255 (65.7) | 100 (74.9)
Statistical Analysis 1: Comparison: Epanova 4 g vs Lovaza 4 g; Test type: Superiority or Other; p = 0.0025, Mixed Models Analysis — The p-value was only interpreted descriptively; Geometric mean ratio in % = 298.91, 95% CI 2-sided [164.32 to 543.74]
Statistical Analysis 2: Comparison: Epanova 2 g vs Lovaza 4 g; Test type: Superiority or Other; p = 0.0418, Mixed Models Analysis — The p-value was only interpreted descriptively; Geometric mean ratio in % = 187.28, 95% CI 2-sided [102.95 to 340.66]

5. Secondary Outcome: Baseline-adjusted AUC0-24 for Plasma Total DHA
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ug/mL
Arm/Group | Epanova 2 g | Epanova 4 g | Lovaza 4 g
Number analyzed (Participants) | 6 | 6 | 12
hr*ug/mL | 1710 (136.3) | 1550 (195.2) | 2190 (86.9)
Statistical Analysis 1: Comparison: Epanova 4 g vs Lovaza 4 g; Test type: Superiority or Other; p = 0.6833, Mixed Models Analysis; Geometric mean ratio in % = 79.36, 95% CI 2-sided [22.95 to 274.45]
Statistical Analysis 2: Comparison: Epanova 2 g vs Lovaza 4 g; Test type: Superiority or Other; p = 0.5220, Mixed Models Analysis; Geometric mean ratio in % = 69.39, 95% CI 2-sided [20.07 to 239.98]

6. Secondary Outcome: Baseline-adjusted Cmax for Plasma Total DHA
Time Frame: This is a crossover study with two treatment periods. The estimated treatment effects were based on the within-subject comparison between the two treatments, each having a 4-week duration and a 4-week wash off period in between.
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Epanova 2 g | Epanova 4 g | Lovaza 4 g
Number analyzed (Participants) | 6 | 6 | 12
ug/mL | 116 (76.1) | 118 (89.2) | 128 (82.3)
Statistical Analysis 1: Comparison: Epanova 4 g vs Lovaza 4 g; Test type: Superiority or Other; p = 0.9034, Mixed Models Analysis; Geometric mean ratio in % = 104.78, 95% CI 2-sided [44.92 to 244.41]
Statistical Analysis 2: Comparison: Epanova 2 g vs Lovaza 4 g; Test type: Superiority or Other; p = 0.5782, Mixed Models Analysis; Geometric mean ratio in % = 80.58, 95% CI [34.55 to 187.95]

7. Secondary Outcome: Baseline-adjusted AUC0-24 for Plasma Total DPA
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ug/mL
Arm/Group | Epanova 2 g | Epanova 4 g | Lovaza 4 g
Number analyzed (Participants) | 6 | 6 | 12
hr*ug/mL | 244 (225.3) | 380 (240.9) | 108 (374.3)
Statistical Analysis 1: Comparison: Epanova 4 g vs Lovaza 4 g; Test type: Superiority or Other; p = 0.0391, Mixed Models Analysis; Geometric mean ratio in % = 753.75, 95% CI 2-sided [112.03 to 5071.6]
Statistical Analysis 2: Comparison: Epanova 2 g vs Lovaza 4 g; Test type: Superiority or Other; p = 0.9578, Mixed Models Analysis; Geometric mean ratio in % = 104.98, 95% CI 2-sided [15.60 to 706.33]

8. Secondary Outcome: Baseline-adjusted Cmax for Plasma Total DPA
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Epanova 2 g | Epanova 4 g | Lovaza 4 g
Number analyzed (Participants) | 6 | 6 | 12
ug/mL | 23.0 (64.2) | 26.4 (83.3) | 11.1 (128.9)
Statistical Analysis 1: Comparison: Epanova 4 g vs Lovaza 4 g; Test type: Superiority or Other; p = 0.0186, Mixed Models Analysis; Geometric mean ratio in % = 376.64, 95% CI 2-sided [128.55 to 1103.5]
Statistical Analysis 2: Comparison: Epanova 2 g vs Lovaza 4 g; Test type: Superiority or Other; p = 0.5955, Mixed Models Analysis; Geometric mean ratio in % = 131.74, 95% CI 2-sided [44.97 to 386.00]

ADVERSE EVENTS:
Groups:
- Epanova 2 g (I); Epanova 4 g (I); Lovaza 4 g (I): Treatment period I
- Epanova 2 g (II); Epanova 4 g (II); Lovaza 4 g (II): Treatment period II
Arm/Group | Epanova 2 g (I) | Epanova 4 g (I) | Lovaza 4 g (I) | Epanova 2 g (II) | Epanova 4 g (II) | Lovaza 4 g (II)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/8 | 0/4 | 0/2 | 0/7
Other Adverse Events (participants affected / at risk) | 2/3 | 3/4 | 5/8 | 3/4 | 2/2 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epanova 2 g (I) (N=3) | Epanova 4 g (I) (N=4) | Lovaza 4 g (I) (N=8) | Epanova 2 g (II) (N=4) | Epanova 4 g (II) (N=2) | Lovaza 4 g (II) (N=7)
Any (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Any (Gastrointestinal disorders) | 2 | 2 | 2 | 2 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Any (General disorders) | 0 | 1 | 3 | 2 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Any (Infections and infestations) | 1 | 2 | 0 | 1 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Any (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Any (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Any (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Any (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Any (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Xanthelasma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Xanthoma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No